CLINICAL TRIAL: NCT04791696
Title: Risk Factors for Human Corneal Graft Failure : a Monocentric Retrospective Observational Cohort, Montpellier, South of France
Brief Title: Risk Factors for Human Corneal Graft Failure : a Monocentric Retrospective Observational Cohort
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0148
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Corneal Transplant Rejection
Keywords: Cornea / surgery; Corneal Transplantation* / adverse effects; Corneal Transplantation* / methods; Graft Rejection / prevention & control; Humans
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Keratoplasty is one of the most common grafts and penetrating keratoplasty is still the technique most used in the world, ahead of lamellar grafts, and is estimated to represent 70% of the total.

Graft rejection is still the main cause of failure of this type of surgery, to the extent that nearly a third of all patients will in some way be affected by rejection in due course.

Numerous risk factors for rejection have been identified, whether related to the donor, the recipient, or the surgical procedure itself.

In addition, many of the studies performed have used univariate analysis only, and yet there is a strong case for multivariate analysis, given the wide range of factors that need to be examined.

This study seeks to analyze the rejection rates and the survival of penetrating keratoplasty for a group of patients from Montpellier Hospital (France).

ELIGIBILITY:
Inclusion criteria:

-keratoplasty performed in the ophthalmology department of the CHRU of Montpellier between 15/06/2005 and 18/09/2018

Exclusion criteria:

* a non-optical graft (tectonic and analgesic graft)
* lamellar graft (DALK (Deep Anterior Lamellar Keratoplasty) and DSAEK (Descemet Stripping Automated Endothelial Keratoplasty))
* Silica gel re-dried cornea, duplicates (we included each patient only once per eye)
* medical record missing from the archives.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutives keratoplasty performed in the ophthalmology department of the CHRU (Centre Hospitalier Régional Universitaire) of Montpellier between 15/06/2005 and 18/09/2018, a period of just over 13 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
graft rejection | 1 day
  The main criterion studied is the fact that rejection had occurred, defined by the appearance of a rejection line, whether epithelial or endothelial (Khodadoust line), subepithelial infiltrates, or an anterior chamber inflammatory reaction (Tyndall effect, retro corneal precipitates and Descemet folds) with corneal edema in a previously clear graft. Opaque grafts with no clear period in the 2 weeks after grafting were not considered as rejections, but rather as straightforward graft failures.

SECONDARY OUTCOMES:
irreversible graft rejection | 1 day
  The other criteria studied is irreversible graft rejection, defined as the persistence of a central corneal edema for 3 months despite treatment, and graft failure, defined as a second keratoplasty, or the persistence of a central corneal edema persisting for more than 3 months, whatever the cause (rejection, corneal endothelial cell failure, other).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent DAIEN, MD, PhD, HDR, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Debourdeau E, Builles N, Couderc G, Boulhic J, Chamard C, Villain M, Babeau F, Daien V. Risk factors of rejection after penetrating keratoplasty: a retrospective monocentric study. Graefes Arch Clin Exp Ophthalmol. 2022 Nov;260(11):3627-3638. doi: 10.1007/s00417-022-05691-w. Epub 2022 May 12. PMID 35546638